CLINICAL TRIAL: NCT06358157
Title: Evaluation of the Safety and Performance of the Ladera Medical Suture-Mediated Large Bore Closure (LBC) System
Brief Title: The Ladera Large Bore Closure Feasibility Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ladera Medical (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN02001
Record Dates: First submitted 2024-03-29; First posted 2024-04-10 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Vascular Closure; Femoral Arteriotomy Closure

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Ladera LBC System (Experimental): The Ladera LBC System will be used in all participants enrolled in the study
  Interventions: Device: Ladera LBC System

INTERVENTIONS:
Device: Ladera LBC System — Use of the Ladera LBC System to close the femoral arteriotomy

SUMMARY:
This study evaluates the safety and performance of the Ladera Medical suture-mediated large bore closure (LBC) system in gaining post procedure hemostasis in subjects undergoing interventional catheterization procedures using a large-bore procedure sheath.

DETAILED DESCRIPTION:
The Ladera Medical suture mediated large bore closure (LBC) system is a vascular closure device intended for use in catheterization laboratories following percutaneous interventional catheterization procedures that use the retrograde common femoral artery access route for large bore interventional devices. The function of Ladera LBC System is to percutaneously close the puncture in the artery wall (arteriotomy) through which the catheters were inserted for the procedure.

The study is being conducted to demonstrate the safety and performance of the LBC System in achieving hemostasis in femoral arterial access sites in subjects undergoing percutaneous interventional catheterization procedures using a large-bore procedure sheath.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 or older
2. Scheduled for an elective or planned single percutaneous interventional catheterization procedure involving access through the femoral artery using a unilateral procedural sheath ID within the indicated range or device (OD) if an expandable sheath is used
3. Willing and able to give written informed consent and to complete a follow-up visit at 30 ± 7 days

Exclusion Criteria:

Baseline

1. Evidence of current systemic bacterial or cutaneous infection, including groin infection
2. Known bleeding disorders including thrombocytopenia (platelet count < 100,000), thrombasthenia, hemophilia or Von Willebrand's disease or known Type II heparin-induced thrombocytopenia
3. Thrombolytics (e.g., streptokinase, urokinase), Angiomax (bivalirudin) or other thrombin-specific anticoagulants planned within 24 hours prior to primary procedure
4. Glycoprotein IIb/IIIa inhibitors planned within 24 hours prior to the primary procedure, during the procedure, or within 48 hours after the primary procedure
5. Planned anticoagulation therapy within 24 hours after the primary procedure such that the activated clotting time (ACT) is expected to be elevated greater than 250 seconds
6. Significant anemia (hemoglobin less than 9 g/dL or hematocrit less than 27%)
7. Significant blood loss requiring transfusion of blood products within 30 days prior to primary procedure
8. Documented left ventricular ejection fraction less than 20%
9. Renal insufficiency (glomerular filtration rate less than 30 ml/min or baseline serum creatinine greater than 2.5 mg/dL) or on renal replacement therapy
10. Significant inflow disease (iliac or artery diameter stenosis greater than 50%) and/or severe peripheral arterial disease (Rutherford Category 5 or 6), as confirmed with pre-primary procedure CT angiography
11. Common femoral artery lumen diameter less than the indicated minimum based on pre-primary procedure CT angiography
12. Evidence of marked tortuosity of the femoral or external iliac arteries in the target leg, based on pre-primary procedure CT angiography
13. Evidence of arterial diameter stenosis (greater than 30%) within 15 mm proximal or distal to arteriotomy site based on pre-primary procedure CT angiography
14. Evidence of anterior wall calcification of the target common femoral artery (other than small, diffuse deposits which in the opinion of the Investigator will not impede the vascular closure procedure) within 15 mm proximal or distal to arteriotomy site based on pre-primary procedure CT angiography
15. Prior target artery closure with any closure device within 90 days prior to the primary procedure, or closure with manual/mechanical compression within 30 days prior to the primary procedure
16. Prior atherectomy, stent, vascular surgery, or vascular graph in the common femoral artery of target leg
17. Known existing nerve damage in the target leg
18. Unsuitable for surgical repair of the target leg access site
19. Connective tissue disease (e.g., Marfan's Syndrome), or significant scarring of the target access site which in opinion of the Investigator, would preclude use of the investigational device in accordance with the IFU
20. Recent (within 60 days) cerebrovascular accident or Q-wave myocardial infarction
21. Morbidly obese or cachectic (BMI greater than 40 kg/m2 or less than 20 kg/m2)
22. Planned major intervention or surgery, including planned endovascular/catheter-based procedure, in the target leg in the 30 days following the primary procedure
23. Ipsilateral or contralateral lower extremity amputation
24. Non-ambulatory (confined to bed or wheelchair)
25. Known allergy to any of the materials used in the LBC System (refer to Instructions for Use)
26. Pregnant, lactating, or planning to become pregnant within 30 days following the primary procedure
27. Would refuse blood transfusion if it were to be needed
28. Current enrollment in another investigational medical device or drug study
29. Previous participation in this study
30. Other medical, social, or psychiatric condition that in the opinion of the Investigator would interfere with participation in the study

Intra-Procedural

1. Access site tissue tract (i.e., estimated distance from skin entry point to arterial anterior surface at arteriotomy) expected to be greater than the indicated maximum
2. Initial common femoral arterial access for the primary procedure achieved with manual palpation or blind arterial stick access, without use of an image guided approach (ultrasound or angiography)
3. During arterial puncture for the primary procedure, the target femoral artery suspected to have experienced a posterior arterial wall needle puncture or need for greater than 2 ipsilateral arterial punctures
4. Primary procedural access site in the profunda femoris or superficial femoral artery or the bifurcation of these vessels
5. Primary procedural access site located at the level or above the inferior epigastric artery and/or above the inguinal ligament based on bony/arterial landmarks (above femoral head on A-P projection)
6. Difficult dilation during initial target femoral artery access (e.g., that damages or kinks dilators) while step-dilating up to the primary procedural sheath
7. Primary procedural access site is in a vascular graft
8. Primary procedural sheath ID greater than the indicated size, or primary procedural device greater than the indicated size if an expandable sheath is used
9. Significant blood loss requiring transfusion of blood products during primary procedure
10. Evidence of overt, actionable bleeding around the primary procedure sheath
11. Primary procedure sheath in place longer than 6 hours
12. Evidence of an acute hematoma (greater than 2 cm in diameter), arteriovenous fistula, pseudoaneurysm, or intraluminal thrombosis at the primary procedure access site
13. Angiographic evidence of laceration, dissection or stenosis in the femoral artery that would preclude use of the investigational device
14. Ipsilateral femoral venous sheath during the primary procedure
15. Activated clotting time (ACT) greater than the target immediately prior to primary sheath removal and planned vascular closure or if ACT measurements are expected to be greater than the target seconds within 24 hours after primary procedure
16. Uncontrolled hypertension (systolic blood pressure greater than the systolic maximum or diastolic blood pressure greater than the diastolic maximum) at the time of primary sheath removal and planned vascular closure
17. Systolic blood pressure less than the systolic minimum at the time of primary procedural sheath removal and planned vascular closure

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint: Major Arterial Access Site Closure-related Complications | Through 30 days post-procedure
  Assessment of the incidence of major adverse events of the target limb access site through 30 days post procedure attributed directly to the use of the Ladera LBC System without other likely cause analyzed on a per-participant basis.
Primary Performance Endpoint: Time to Hemostasis | Post-procedure, usually within 3 hours
  Elapsed time (min) from the removal of the Ladera LBC System and the primary procedural guidewire to first observed cessation of common femoral artery (CFA) bleeding, excluding cutaneous or subcutaneous oozing that is controlled with light/non-occlusive manual or mechanical pressure, and in the absence of a developing hematoma

SECONDARY OUTCOMES:
Secondary Safety Endpoint: Minor Arterial Access Site Closure-related Complications | Through 30 days post-procedure
  Assessment of the incidence of minor complications of the target limb access site through 30 days post procedure attributed directly to the use of the Ladera LBC System without other likely cause analyzed on a per-participant basis.
Secondary Performance Endpoint: Time-to-Ambulation | Post-procedure, usually within 12 hours
  Time (hrs) from access site closure and primary procedural guidewire removal to when the participant stands and walks at least 20 ft/6 m without evidence of re-bleeding from the access site
Secondary Performance Endpoint: Time-to-Discharge Eligibility | Post-procedure, usually within 48 hours
  Elapsed time (hours) from access site closure and primary procedural guidewire removal to when the participant is eligible for discharged from the hospital based on the assessment of the attending physician
Secondary Performance Endpoint: Incidence of Procedural Success | Through 30 days post-procedure
  Incidence of hemostasis with use of the Ladera LBC System without major access site closure related complications
Secondary Performance Endpoint: Incidence of Device Technical Success | Post-Procedure, usually within 3 hours
  Incidence of successful deployment of the Ladera LBC System and achievement of hemostasis

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Macquarie University, Sydney, New South Wales
  - Alfred Health, Melbourne, Victoria
  - Monash Health, Victoria Heart Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No